CLINICAL TRIAL: NCT04343274
Title: Expanded Access for BLZ-100 (Tozuleristide)
Status: No longer available | Type: Expanded Access
Sponsor: Blaze Bioscience Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BLZ-100EA
Record Dates: First submitted 2020-04-09; First posted 2020-04-13 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

MeSH Terms: interventions — tozuleristide

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Tozuleristide
  Other Names: BLZ-100; Tumor Paint

SUMMARY:
This is the Blaze Bioscience expanded access program for its investigational drug tozuleristide intended for patients with life-threatening diseases or conditions who have exhausted approved treatment options and are unable to participate in a clinical trial involving the investigational drug tozuleristide.

DETAILED DESCRIPTION:
1. Contact Information: A licensed treating physician may submit questions or requests on behalf of a patient regarding expanded access to tozuleristide to be evaluated in accordance with Blaze Bioscience company policies. Physician Expanded Access Requests should be submitted in writing to expandedaccess@blazebioscience.com and include "Expanded Access Request" in the subject.
2. Request Procedures:

   1. General Criteria: Blaze Bioscience will evaluate and respond to each Expanded Access Request individually and on a case-by-case basis. Criteria Blaze Bioscience will use in its evaluation of whether to grant Expanded Access Request include:

      1. Adequate supply of the investigational drug tozuleristide must be available above and beyond the supply needed for Blaze Bioscience clinical trials;
      2. There is sufficient clinical data to identify an appropriate dose of the investigational drug;
      3. There is a good understanding of the patient's clinical situation and investigational drug proposed use for surgery including the proposed fluorescence detection device;
      4. All available therapeutic approaches for the patient's disease have been exhausted by the patient and their physicians;
      5. The investigational drug is considered an "eligible investigational drug" under Section 561(B)(2) of the FDCA at the time of the Expanded Access Request;
      6. Providing the investigational drug is compliant with all applicable rules and laws;
      7. Appropriate Institutional Review Board/Ethics Committee and FDA authorization requested expanded access has been obtained;
      8. Treating physician understands and is willing to be responsible for ensuring that the patient informed consent requirements are met; and
      9. Treating physician understands and is willing to be the holder of a treatment IND with FDA.
   2. Timing of acknowledgement: Blaze Bioscience endeavors to acknowledge requests within ten (10) business days of receipt of an Expanded Access Request.
   3. Clinical trials: Blaze Bioscience lists its active clinical trials on clinicaltrials.gov. Before granting an Expanded Access Request for tozuleristide, written confirmation by the treating physician that the patient is not eligible for an active Company clinical trial is needed prior to consideration of the Expanded Access Request.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing surgery for suspected or confirmed tumor
* Not eligible for current clinical trials of tozuleristide

Age Groups: Child, Adult, Older Adult